CLINICAL TRIAL: NCT05814510
Title: Implementation of Asthma Community Home and School Management Program (Asthma CHAMPS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Baltimore City Public Schools (Unknown); Baltimore City Health Department (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB00301358; HL157845 (Other: NHLBI)
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- School staff (Experimental): School staff in a K-8 school participating in Asthma CHAMPS
  Interventions: Behavioral: Asthma CHAMPS full program; Behavioral: Asthma CHAMPS Wait List Control
- Children with asthma (Experimental): Aged 5-13 and enrolled in Baltimore City Public School participating in Asthma CHAMPS
  Interventions: Behavioral: Asthma CHAMPS full program; Behavioral: Asthma CHAMPS Wait List Control
- Caregivers of children with asthma (Experimental): Caregiver of a child with asthma that is aged 5-13 enrolled in a Baltimore City Public School participating in Asthma CHAMPS
  Interventions: Behavioral: Asthma CHAMPS full program; Behavioral: Asthma CHAMPS Wait List Control

INTERVENTIONS:
Behavioral: Asthma CHAMPS full program — Full program includes (1) education for staff, students, and caregivers (2) environmental education and intervention (3) asthma care coordination (4) resources
Behavioral: Asthma CHAMPS Wait List Control — Stepped wedge design

SUMMARY:
The long-term goal is to implement an evidence-based asthma intervention based on the Center for Disease Control's recommended framework (EXHALE) within Baltimore City Public Schools (BCPS). As part of a stepped wedge pragmatic trial the investigators will:

1. Evaluate the effectiveness of a tailored implementation plan of Asthma CHAMPS in 32 Baltimore city elementary schools to reduce asthma disparities.
2. Conduct a pragmatic trail using a stepped wedge design to evaluate implementation of a school and home asthma intervention program to reduce asthma-related absences, healthcare utilization and exacerbations and improve asthma control, among children enrolled in 32 Baltimore City elementary schools.
3. Use qualitative methods (observation and semi structured interviews) to obtain stakeholder feedback (parents, community health workers, school personnel and administrators) on impact of Asthma CHAMPS, identify potential refinements in intervention and implementation strategies, and evaluate impact of local adaptation and fidelity on implementation success and sustainability.

DETAILED DESCRIPTION:
Implementation Aim: Evaluate the effectiveness of a tailored implementation plan of Asthma CHAMPS in 32 Baltimore city elementary schools to reduce asthma disparities.

Hypothesis: The investigators hypothesize that Baltimore City schools will have greater adoption and penetration of Asthma CHAMPS (e.g. more schools participating, and more staff and family asthma education sessions), greater feasibility/acceptability (e.g. more staff participating in asthma care activities, greater staff confidence in managing asthma) and greater satisfaction and appropriateness with a tailored implementation strategy compared to wait list-control group.

The long-term goal is to implement an evidence-based asthma intervention based on the Centers for Disease Control (CDC) recommended framework (EXHALE)14 within BCPS. To provide the foundation for success, the investigators will identify and engage local key stakeholders, conduct a community needs assessment to inform necessary refinement and adaptations of the interventions, and develop a tailored collaborative strategy to ensure successful implementation of an asthma intervention program. Results for this multi-phase project will identify best practices for implementation of a tailored multi-level asthma intervention program (Asthma CHAMPS: Community and Home Asthma Management Program in Schools), within Baltimore City Schools to reduce asthma disparities.

Effectiveness Aim: Conduct a pragmatic trail using a stepped wedge design to evaluate implementation of a school and home asthma intervention program to reduce asthma-related absences, healthcare utilization and exacerbations and improve asthma control, among children enrolled in 32 Baltimore City elementary schools.

Hypothesis: Children with asthma who attend schools engaged in Asthma CHAMPS program will have improved asthma outcomes, including improved asthma control, reduced ED visits/hospitalizations and courses of oral corticosteroids and impact (reduced asthma-related school absences).

Qualitative Aim: Use qualitative methods (observation and semi structured interviews) to obtain stakeholder feedback (parents, community health workers, school personnel and administrators) on impact of Asthma CHAMPS, identify potential refinements in intervention and implementation strategies, and evaluate impact of local adaptation and fidelity on implementation success and sustainability.

ELIGIBILITY:
Adult

Inclusion Criteria:

* Aged 18 or older
* Current caregiver of child with asthma or staff member at a Baltimore City K-8 Public School in Asthma CHAMPS

Exclusion Criteria:

* Unwilling to consent

Children with asthma

Inclusion Criteria:

* Asthma diagnosis
* Currently enrolled in Baltimore City K-8 Public School participating in Asthma CHAMPS

Exclusion Criteria:

* Unwilling to provide assent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Asthma-related absences | 4 years
  Administrative data from schools on attendance for child with asthma
Emergency Department (ED) utilization for asthma by children | 4 years
  Counts of ED visits for asthma
Hospitalization for asthma by children | 4 years
  Counts of hospital admissions for asthma
Oral corticosteroid steroid prescription for asthma by children | 4 years
  Counts of prescribed oral corticosteroids for asthma

SECONDARY OUTCOMES:
Intervention penetration as assessed by counts | 4 years
  Counts of asthma education sessions for family and staff
Acceptability of Intervention (AIM) as assessed by a 4 item questionnaire | 4 years
  4 item measure of implementation outcome often considered "leading indicator" of implementation success. Administered on a 5 point Likert scale with higher scores indicating greater agreement with specific items.
Intervention Appropriateness Measure (IAM) as assessed by a 4 item questionnaire | 4 years
  4 item measure of implementation outcome often considered "leading indicator" of implementation success. Administered on a 5 point Likert scale with higher scores indicating greater agreement with specific items.
Feasibility of Intervention (FIM) as assessed by a 4 item questionnaire | 4 years
  4 item measure of implementation outcome often considered "leading indicator" of implementation success. Administered on a 5 point Likert scale with higher scores indicating greater agreement with specific items.
Intervention Satisfaction as assessed by a composite measure | 4 years
  Composite measure administered to staff and caregivers with items assessing asthma management motivation and confidence. Answer options are on a scale of 1-10 with higher scores generally indicating greater agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle N Ealin, PhD, Principal Investigator — JHU; Meredith McCormack, MD MHS, Principal Investigator — JHU
Locations (1):
- Baltimore City Public Schools, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No